CLINICAL TRIAL: NCT00988273
Title: Confocal Endomicroscopy in Patients Undergoing Endoscopy
Brief Title: Confocal Endomicroscopy During Endoscopy
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: 20090821300
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2012-04

CONDITIONS: Inflammatory Bowel Disease
Keywords: Crohn's disease; Ulcerative colitis; dysplasia
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: In patients undergoing endoscopy for indications other than Crohn's disease or ulcerative colitis
  Interventions: Device: Confocal endomicroscopy
- Diseased group: Patients with Crohn's disease or ulcerative colitis undergoing endoscopy.
  Interventions: Device: Confocal endomicroscopy

INTERVENTIONS:
Device: Confocal endomicroscopy — Patients will undergo confocal endomicroscopy during their endoscopy, and findings of the confocal endomicroscopy in the control group will be compared to the diseased group.
  Other Names: laser confocal endomicroscopy
  Groups: Control
Device: Confocal endomicroscopy — Patients will undergo confocal endomicroscopy during their endoscopy, and findings of the confocal endomicroscopy in the diseased group will be compared to the control.
  Other Names: laser confocal endomicroscopy
  Groups: Diseased group

SUMMARY:
The main objective of this study is to determine the role of epithelial cell homeostasis in the pathogenesis of intestinal diseases.

Background: Alterations in intestinal barrier function may play a significant role in the pathogenesis of chronic intestinal diseases such as inflammatory bowel disease (IBD). The intestinal epithelium functions as a barrier to the luminal contents, thereby preventing undesirable solutes, micro-organisms and other luminal antigens from entering the body. Confocal endomicroscopy has recently been shown that increased epithelial cell shedding may contribute to increased intestinal permeability, at least locally. In our study, we want to determine the contribution of epithelial cell shedding to intestinal permeability in vivo in patients with inflammatory bowel disease compared to controls.

Scope:

In inflammatory bowel disease patients and controls (patients undergoing endoscopy for other indications).

Methods:

We will perform confocal endoscopy during the patient's endoscopic procedure.

Procedure:

The patient will receive intravenous fluorescein, followed by confocal imaging of the gastrointestinal tissue. The images are captured on the computer. The proposed study will provide important insights into epithelial cell shedding as a contributor to altered intestinal permeability.

ELIGIBILITY:
Inclusion Criteria for patients includes:

1. Subjects over 18 years of age.
2. Subjects undergoing endoscopic procedures such as gastroscopy, colonoscopy, endoscopic retrograde cholangiopancreatography and endoscopic ultrasound will all be included.

Exclusion Criteria:

1. Under 18 years of age.
2. Cognitively impaired.
3. Residing in institutions (eg. prison, extended care facility)
4. Employees of research(s)' organization
5. In emergency or life-threatening situations
6. Have language barriers (eg. illiterate, not English-speaking, dysphasic) preventing adequate consent process
7. Resides in another country

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing endoscopy: study group are patients evaluated for IBD symptoms and control patients for other indications such as colon cancer screening, positive fecal occult testing, constipation or diarrhea.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2009-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The intestinal morphology as visualized using confocal laser endomicroscopy | 3 years.
  Intestinal morphology as measured by epithelial cells and gaps, presence of bacteria in the epithelial lining and the lamina propria will be quantitated.

SECONDARY OUTCOMES:
Clinical outcome and pathologic/molecular correlation with intestinal morphology | 3 years.
  The clinical outcomes of inflammatory bowel patients, location and severity of their disease, and correlation with molecular studies including tissue cytokine levels will be studied.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Liu JJ, Wong K, Thiesen AL, Mah SJ, Dieleman LA, Claggett B, Saltzman JR, Fedorak RN. Increased epithelial gaps in the small intestines of patients with inflammatory bowel disease: density matters. Gastrointest Endosc. 2011 Jun;73(6):1174-80. doi: 10.1016/j.gie.2011.01.018. Epub 2011 Mar 11. PMID 21396639
- [Background] Turcotte JF, Wong K, Mah SJ, Dieleman LA, Kao D, Kroeker K, Claggett B, Saltzman JR, Wine E, Fedorak RN, Liu JJ. Increased epithelial gaps in the small intestine are predictive of hospitalization and surgery in patients with inflammatory bowel disease. Clin Transl Gastroenterol. 2012 Jul 26;3(7):e19. doi: 10.1038/ctg.2012.13. PMID 23238291
- [Background] Liu JJ, Davis EM, Wine E, Lou Y, Rudzinski JK, Alipour M, Boulanger P, Thiesen AL, Sergi C, Fedorak RN, Muruve D, Madsen KL, Irvin RT. Epithelial cell extrusion leads to breaches in the intestinal epithelium. Inflamm Bowel Dis. 2013 Apr;19(5):912-21. doi: 10.1097/MIB.0b013e3182807600. PMID 23511029
- [Background] Turcotte JF, Kao D, Mah SJ, Claggett B, Saltzman JR, Fedorak RN, Liu JJ. Breaks in the wall: increased gaps in the intestinal epithelium of irritable bowel syndrome patients identified by confocal laser endomicroscopy (with videos). Gastrointest Endosc. 2013 Apr;77(4):624-30. doi: 10.1016/j.gie.2012.11.006. Epub 2013 Jan 26. PMID 23357497